CLINICAL TRIAL: NCT02327234
Title: Assessment of Repeated Allergen Challenge and the Effects of Ibuprofen on the Inflammatory Process
Brief Title: Airway Response to Repeat Allergen Challenge and the Effect of Ibuprofen in Mild Atopic Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Don Cockcroft, Professor, University of Saskatchewan
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: Bio REB 14-283
Record Dates: First submitted 2014-12-17; First posted 2014-12-30 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Atopic Asthma
MeSH Terms: interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ibuprofen (Experimental): 400mg (2X200mg) ibuprofen single dose once
  Interventions: Drug: ibuprofen
- Placebo (Placebo Comparator): identical appearing lactose capsules single dose 2 capsules once
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ibuprofen — 2x 200mg ibuprofen, single dose, blinded in 00 capsules
  Other Names: Advil
  Arms: Ibuprofen
Drug: Placebo — lactose filled 00 capsules to match appearance of ibuprofen intervention
  Arms: Placebo

SUMMARY:
The study will assess airway responses in mild atopic asthmatics undergoing repeat allergen challenge testing and will investigate whether ibuprofen changes the response.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of mild asthma, currently well controlled requiring only a bronchodilator (e.g. salbutamol) as needed and infrequently
* has allergies that trigger asthma
* responds to methacholine challenge at 16mg/ml or less
* has FEV1 > 69.5% predicted

Exclusion Criteria:

* respiratory illness within 4 weeks
* other medical condition assessed by the principal investigator that would put the participant at risk or influence the integrity of the data
* pregnant or lactating females
* hypersensitivity to ibuprofen

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Airway response to inhaled allergen | at time of allergen inhalation challenge and for 7 hours after
  area under forced expiratory volume in one second versus time curve; 0-3hours (early response) and 3-7 hours (late response)

SECONDARY OUTCOMES:
Airway response to inhaled methacholine | day before allergen inhalation challenge and 8 hours after allergen inhalation challenge
  delta log methacholine PC20 (provocative concentration of methacholine causing a 20% decrease in the forced expiratory volume in one second)

CONTACTS AND LOCATIONS:
Overall Officials: Don Cockcroft, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: Yes
journal publication

REFERENCES:
- [Derived] Nomani S, Cockcroft DW, Davis BE. Allergen inhalation challenge, refractoriness and the effects of ibuprofen. Allergy Asthma Clin Immunol. 2016 May 24;12:24. doi: 10.1186/s13223-016-0127-z. eCollection 2016. PMID 27222654